CLINICAL TRIAL: NCT06191809
Title: Evaluate the Effectiveness of Progestin-Primed Versus GnRH Antagonist Protocols in Vietnamese Women Undergoing In-vitro Fertilization: A Randomized Controlled Trial
Brief Title: Evaluate the Effectiveness of Progestin-Primed Versus GnRH Antagonist Protocols in Vietnamese Women Undergoing In-vitro Fertilization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Thach Than Trong, Principal Investigator, Hanoi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9720105
Record Dates: First submitted 2023-12-16; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: IVF
Keywords: ppos protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPOS protocol (Active Comparator): Ovarian stimulation protocol used progestin as premature LH surge inhibitor
  Interventions: Procedure: Controlled Ovarian Stimulation Protocol
- GnRH-ant protocol (Active Comparator): Ovarian stimulation protocol used GnRH antagonist as premature LH surge inhibitor
  Interventions: Procedure: Controlled Ovarian Stimulation Protocol

INTERVENTIONS:
Procedure: Controlled Ovarian Stimulation Protocol — Ovarian Stimulation Process:
  * Stimulate ovaries with FSH & hMG (150-375 IU) starting day 2-3 of menstruation.
  * Monitor response with ultrasound & hormones (E2, LH, P4).
  * GnRH-ant arm: Prevent LH surge with Cetrorelix (0.25mg) starting day 5.
  * PPOS arm: Suppress LH with Dydrogesterone (10mg x 3/day) from day 1.
  * Trigger ovulation when ≥2 follicles >17mm (Triptorelin, hCG, or rhCG).
  * Oocyte retrieval 36-38 hours later (>10mm follicles aspirated).
  Embryo Culture & Monitoring:
  * Fertilize with ICSI.
  * Culture & evaluate embryos (43-45 hours, day 3/5).
  * Freeze all embryos.

SUMMARY:
This study aims to evaluate the efficacy of the progestin-primed ovary stimulation (PPOS) protocol compared to the standard GnRH antagonist (GnRH_ant) protocol across successive stages in a controlled ovarian stimulation (COS) and ICSI procedure.

DETAILED DESCRIPTION:
Materials and Method

This was an open-label, randomized controlled trial conducted at the Assisted Reproduction Center of Tam Anh General Hospital. The study aimed to estimate the efficacy of the intervention (PPOS protocol) compared to a control group receiving a gonadotropin-releasing hormone (GnRH) antagonist protocol.

Sample size estimation

The sample size estimation procedure is detailed in the study protocol. In brief, the investigators conducted a simulation that implied the method by Cundill and Alexander (2015) with parameters derived from the clinical profile of 804 patients who underwent ovarian stimulation by two protocols at Tam Anh Hospital from January to October 2022. The procedure aimed to optimize non-inferiority testing on the difference in the quantity of retrieved oocytes between two groups, estimated by a Negative Binomial distribution. The simulation result indicated that a total sample size of 200 patients (n=100 for each treatment arm) would be required to achieve a statistical power of 0.8.

Recruitment of study participants

Infertile patients come for examination at the Assisted Reproduction Center of Tam Anh General Hospital, Hanoi, and the Assisted Reproduction and Graft Technology Center of Hanoi Medical University. In the basic infertility examination process at the hospital, the clinicians will consider the patient's inclusive and exclusive criteria. The clinicians will contact a research team member if the inclusive criteria are met. A research team member or hospital physician will invite the patient to participate, advise on the study procedure and the benefits and risks of participating, and answer any patient questions. If the patients agree to participate, they will consent to participate in the trial. Each participant will be randomly assigned to the treatment group using the PPOS protocol or the control group using the GnRH-ant regimen.

Treatment method

Ovarian stimulation protocols

Controlled ovarian hyperstimulation commenced on the second day of the menses utilizing recombinant follicle-stimulating hormone. In the gonadotropin-releasing hormone (GnRH) antagonist protocol group, pituitary suppression began on stimulation day six via daily 0.25 milligram GnRH antagonist administration (ganirelix or cetrorelix). In the progestin-primed ovarian stimulation (PPOS) group, 30mg/day of dydrogesterone was initiated on cycle day 2 through to trigger day.

Laboratory protocol

Oocyte-cumulus complexes were incubated for 2 hours in G-IVF medium (Vitrolife) using Origio benchtop incubators to complete nuclear maturation. After removing cumulus cells, denuded oocytes were evaluated under an inverted microscope to validate the achievement of metaphase II status, while degenerate, large, or severely dysmorphic oocytes were excluded. Intracytoplasmic sperm injection (ICSI) was executed 3-4 hours post-retrieval by experienced embryologists. Resultant zygotes were cultured in continuous single media (Fujifilm Irvine Scientific) within tri-gas incubators (37°C, 5% O2, 6% CO2) until day 3. Strict morphological criteria were enforced, only retaining normally fertilized two pronuclei zygotes while eliminating abnormal multinuclear embryos. Cleavage-stage quality was graded at 67-69 hours per Istanbul consensus based on cell number, fragmentation, multinucleation, and uniformity. On post-ICSI day 3, embryologists counseled patients on pursuing blastocyst culture versus cryopreservation. The morphology of the blastocysts was evaluated using the Gardner and Schoolcraft grading system, and embryos meeting the criteria of 3-6 AA/AB/BA blastocysts or 1-2 AA/AB embryos were classified as good quality.

ELIGIBILITY:
Inclusion Criteria:

Women meeting the sample selection criteria are as follows:

* Women age 20 to 45 years old.
* Infertility due to male factors, fallopian tube factors, or unknown causes.
* Undergoing IVF in one COS cycle and intended to apply either GnRH antagonist protocol or PPOS protocol
* Voluntary participation in research.

Exclusion Criteria:

* Any contraindications to ovarian stimulation and IVF/ICSI treatment
* Hyperprolactinemia or other endocrine diseases.
* Those who took hormone drugs within the past 3 months
* Suffering from systemic diseases such as kidney failure, lupus erythematosus, depression, etc.
* Abnormal structure of the uterine cavity.
* Patients with endometriosis or cancer
* Random-start cycles.
* Oocyte donation cycles
* Perform embryo biopsy.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The quantity of day 3rd and day 5th embryos and MII oocytes | 11 months after initiation of treatment in either arm

CONTACTS AND LOCATIONS:
Overall Officials: Thach Than Trong, Principal Investigator — Hanoi Medical University
Locations (1):
- Univesity of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT06191809/Prot_SAP_ICF_000.pdf